CLINICAL TRIAL: NCT04883060
Title: Pilot Testing for Midline Measuring Device
Acronym: MMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Matthew Howard, Professor of Neurosurgery, Head of Department of Neurosurgery at University of Iowa, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201704798
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Ventriculo-Peritoneal Shunt Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Patients undergoing ventriculoperitoneal surgery where the midline localizer was used
  Interventions: Device: midline localizer

INTERVENTIONS:
Device: midline localizer — a midline localizer device with a laser pointer is used to localize where the midline is likely to be located on the patient head prior to the surgery.

SUMMARY:
Identifying the exact middling on the patient's head during the planning phase of surgery is crucial yet can be challenged by patient's head position and hair. The investigators have invented a device that uses anatomical landmark to quickly and gracefully identify the midline on a patient's head. The device is a U-shaped instrument equipped with a laser pointer at the midline. The instrument also has smooth spheres that can be positioned over the patients' ears bilaterally. The midline laser pointer will identify the midline on the patients' head. this measurement procedure is typically done after the patient is placed under anesthesia. The standard way of determining the midline on the skull is simply by surgeon's vision without any measurements. This new technique will be contrasted against the standard way. The device was invented by investigators in neurosurgery (led by Dr. Matthew Howard III). This is not patented it at this time. There is no company involved in manufacturing (assembly was completed with the help of the hospital's machine shop).

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal pressure hydrocephalus who are scheduled to undergo a ventriculoperitoneal shunt surgery

Exclusion Criteria:

* Patients who are not able to consent

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Midline Localization
Description: The average distance separating the staple from the lateral edge of the sagittal sinus
Time Frame: Immediate postop, an average of 4 hours
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intervention
Number analyzed (Participants) | 40
mm | 0.9 (1.6)

2. Secondary Outcome: Burr Hole Placement
Description: Number of participants in which their Burr hole placement was between 3 and 4 cm away from anatomical midline
Time Frame: Immediately Post-op, an average of 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 40
Participants | 37

ADVERSE EVENTS:
Time Frame: From the start of surgery until surgical closure, up to 2.5 hours
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 4/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=40)
Incorrect Burr Hole Placement (Surgical and medical procedures) | 3 (3) — Burr hole was not between 3 and 4 cm away from anatomical midline
Ventricle Catheter Misplacement (Surgical and medical procedures) | 1 (1) — Catheter tip entered the parenchyma at the level of gyrus fasciolaris

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT04883060/Prot_SAP_000.pdf